CLINICAL TRIAL: NCT05510544
Title: Efficacy and Safety of Plerixafor in Patients With Poorly Mobilized Lymphoma
Brief Title: Plerixafor for Poorly Mobilized Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YF-PL-001
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm: plerixafor, G-CSF (Experimental): plerixafor in combination with granulocyte colony stimulating factor (G-CSF) for CD34+ HSC mobilization in poorly mobilized lymphoma patients
  Interventions: Drug: Plerixafor,G-CSF

INTERVENTIONS:
Drug: Plerixafor,G-CSF — G-CSF: 10 μg/kg/day, subcutaneously injected, every morning from day 1 to day 8.
  Plerixafor injection: 0.24 mg/kg/day, subcutaneous injection, starting on the 4th day, once a day, up to 4 times in a row. Plerixafor injection and G-CSF administration site should be separated. The interval between plerixafor injection and stem cell collection was 10-11 hours.
  Other Names: plerixafor, G-CSF

SUMMARY:
Autologous hematopoietic stem cell transplantation is one of the effective means of lymphoma treatment, but patients who receive transplantation in the absence of sufficient stem cell numbers have a delay in stem cell engraftment and a markedly increased risk of infection and emergence. Plerixafor injection is a strong and specific antagonist of CXCR4. It can rapidly mobilize stem cells from bone marrow into peripheral blood circulation by blocking the combination of SDF1 and CXCR4. Studies have shown that the simultaneous use of plerixafor injection and G-CSF can collect more hematopoietic stem cells in a certain period of time than cancer patients who use G-CSF alone. This multicenter, open-label, single-arm study was designed to evaluate the efficacy and safety of plerixafor injection for hematopoietic stem cell mobilization in poorly mobilized lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathological examination confirmed lymphoma;
* Age 18 to 70 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Suitable for autologous peripheral blood hematopoietic stem cell transplantation and plan to use autologous peripheral blood hematopoietic stem cell transplantation for treatment, and obtain partial remission (PR) or complete remission (CR) after anti-tumor therapy;
* Negative bone marrow examination within 45 days (the standard is that the results of bone marrow smear, biopsy and flow cytometry are all negative);
* Any one of the conditions for poor mobilization:

  * Poor steady-state mobilization: rest for 3 weeks or more after the last chemotherapy, give G-CSF 10 μg/kg/day, and peripheral blood CD34+ cells <10/μL on the 4th day of G-CSF treatment;

    * Poor chemotherapy mobilization: When chemotherapy + G-CSF is used for mobilization, on the 7th to 10th day after chemotherapy, or the expected white blood cell (WBC) drops to the lowest point, each participating center starts to give G-CSF 10 μg/kg according to the diagnosis and treatment standards. Treatment, until WBC recovered from the lowest point to 4 × 10ˆ9/L (applicable to WBC decreased to <4 × 10ˆ9/L after chemotherapy) or G-CSF treatment on the 4th day (applicable to WBC after chemotherapy failed to drop to <4 ×10ˆ9/L) CD34+ cells in peripheral blood <10/μL;

      * The amount of CD34+ cells collected on the first day of collection is less than 1×10ˆ6/kg;

        * The amount of CD34+ cells collected 2 days before collection is less than 1.5×10ˆ6/kg;
* Informed consent and signed informed consent voluntarily.

Exclusion Criteria:

* suffering from chronic lymphocytic leukemia;
* Hematopoietic stem cell collection has been performed in the past;
* Received autologous or allogeneic hematopoietic stem cell transplantation in the past;
* Received any radio-immunotherapy in the past (including tiimumab or tosilimumab, etc.);
* Received pelvic radiotherapy in the past;
* Major surgery (excluding diagnostic surgery) within 4 weeks before the first study drug administration;
* Have been vaccinated or will be vaccinated with live vaccines within 30 days before the first study drug administration;
* Human immunodeficiency virus (HIV) positive;
* Patients who meet any of the following laboratory criteria:

  * White blood cell (WBC) count ≤2.5×10ˆ9/L;

    * Absolute neutrophil count (ANC) <1.5×10ˆ9/L;

      * Platelet (PLT) count ≤100×10ˆ9/L;

        * Creatinine clearance ≤50mL/min;

          * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin ≥ 2.5 times the upper limit of normal;
* Those with active infection, including unexplained fever (axillary temperature >37.3℃) or those who need antibiotic, antiviral or antifungal treatment within 7 days before the first use of G-CSF;
* are pregnant or breastfeeding;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients achieving ≥2 × 10ˆ6/kg CD34+ HSCs within ≤4 apheresis sessions. | within 4 days

SECONDARY OUTCOMES:
the proportion of patients achieving ≥5 × 106/kg CD34+ HSCs within ≤4 apheresis sessions. | within 4 days
time to collect ≥2 × 106/kg CD34+ HSCs, | at the end of therapy
time to collect ≥5 × 106/kg CD34+ HSCs, | at the end of therapy
The parameters for safety assessment included adverse event (AE), serious AE (SAE) and treatment emergent adverse event (TEAE) | at the end of therapy，7-21 days after mobilization collection

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China